CLINICAL TRIAL: NCT00305578
Title: Memantine Augmentation of Lamotrigine Incomplete Response in Bipolar Depression: A Randomized Placebo Controlled Clinical Trial
Brief Title: Memantine Augmentation of Lamotrigine Incomplete-Response in Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0501-43
Record Dates: First submitted 2005-09-14; First posted 2006-03-22 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-06

CONDITIONS: Bipolar Depression
Keywords: Bipolar; Depression; Incomplete Response
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo daily
  Interventions: Drug: Placebo
- Memantine (Active Comparator): Daily dose Memantine
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Memantine will be given orally. Subjects will be started at a dose of 5 mg for the first week and then increased by 5 mg every week up to a maximum of 20 mg depending on response and tolerance and will be kept at that level for the rest of the study. This is an 8 week study.
  Other Names: Memantine or Namenda
  Arms: Memantine
Drug: Placebo — No active medication, only placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether addition of memantine to bipolar depression patients who have had an incomplete response to lamotrigine (Lamictal) which is frequently used to treat bipolar depression in the clinical setting. At present, memantine is approved for use in the treatment of Alzheimer's disease or dementia, but not for use for the treatment of bipolar depression. Subjects will be asked to participate because they are suffering from bipolar depression associated and have had an inadequate response to lamotrigine. Subjects will have to be on at least 100 mg per day, for at least 4 weeks.

DETAILED DESCRIPTION:
Hypothesis/Objectives:

H1: Lamotrigine inadequate-response patients augmented with memantine for 8 weeks will have significantly greater improvement on the Hamilton Depression Rating Scale (HDRS) and Clinical Global Improvement (CGI) scale compared to patients augmented with placebo.

H2: Lamotrigine inadequate-response patients augmented with memantine for 8 weeks will have significantly greater improvement of scores on the Selective Reminding Test (SRT), the Digit Span Test, the Stroop Test, and Trail Making Test (TMT) than patients augmented with placebo.

Study Population:

We will study 40 bipolar disorder depressed (BDD) outpatients (20 in each arm) recruited from the outpatient Mood Disorders Clinic and by advertisement.

ELIGIBILITY:
Inclusion Criteria:: 1) age 18 - 65; 2) satisfy DSM-IV-TR criteria for Bipolar Disorder and Major Depressive Episode; 3) Lamotrigine Inadequate-Response: Defined as already treated with at least 100 mg of lamotrigine for at least 4 weeks but 17 item HDRS rating > 15; 4) give informed consent as approved by local IRB; 5) if on other antidepressants or mood stabilizers on stable dose for the past 4 weeks.

Exclusion Criteria:1) comorbid psychotic disorder such as schizophrenia or schizoaffective disorder; 2) significant suicidal or homicidal risk; 3) clinically significant medical illness; 4) allergy or intolerance to lamotrigine or memantine; 5) pregnancy, planning to be pregnant or not using adequate contraception; 6) satisfy criteria for substance dependence within 6 months prior to start of the study; and 7) on any medication with significant adverse interaction with either lamotrigine or memantine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-08; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Adult Psychiatric Clinic, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo daily
  Placebo : No active medication, only placebo
- Memantine: Daily dose Memantine
  Memantine : Memantine will be given orally. Subjects will be started at a dose of 5 mg for the first week and then increased by 5 mg every week up to a maximum of 20 mg depending on response and tolerance and will be kept at that level for the rest of the study. This is an 8 week study.
Period: Overall Study
Arm/Group | Placebo | Memantine
Started | 15 | 14
Completed | 12 | 12
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Memantine | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (14) | 38 (15) | 40 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in 17-item Hamilton Depression Rating Scale From Baseline to 8 Weeks (Baseline - 8 Wks)
Description: Scale for measurement of depression severity. Total of scale is used. Total range is from 0 - 50 with higher score signifying higher severity of depression. Outcome measure is change in score from baseline to 8 wks.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 15 | 14
units on a scale | 7 (6) | 9 (7)

ADVERSE EVENTS:
Arm/Group | Placebo | Memantine
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 14/15 | 11/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Memantine (N=14)
somnolence (Nervous system disorders) | 5 (7) | 3 (6)
shakiness (Nervous system disorders) | 1 (2) | 0 (0)
blurred vision (Nervous system disorders) | 0 (0) | 2 (4)
headache (Nervous system disorders) | 4 (6) | 3 (7)
sharper sense of smell (Nervous system disorders) | 0 (0) | 1 (1)
difficulty concentrating (Nervous system disorders) | 0 (0) | 1 (1)
fatigue (Nervous system disorders) | 1 (3) | 1 (1)
muscle twitching (Nervous system disorders) | 0 (0) | 1 (1)
nocturnal sweating (Nervous system disorders) | 0 (0) | 1 (8)
muscle weakness and muscle spasms (Nervous system disorders) | 1 (1) | 1 (2)
dizziness (Nervous system disorders) | 1 (3) | 1 (1)
dry mouth (Nervous system disorders) | 3 (4) | 1 (3)
insomnia (Nervous system disorders) | 1 (1) | 0 (0)
restlessness (Nervous system disorders) | 1 (4) | 0 (0)
crawling skin (Nervous system disorders) | 1 (2) | 0 (0)
feeling hot (Nervous system disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
gas (Gastrointestinal disorders) | 1 (1) | 1 (1)
indigestion (Gastrointestinal disorders) | 1 (4) | 2 (3)
constipation (Gastrointestinal disorders) | 1 (1) | 1 (2)
diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (4)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
decreased appetite (Gastrointestinal disorders) | 0 (0) | 1 (7)
chest pain and chest tightness, (Cardiac disorders) | 2 (5) | 1 (1)
high blood pressure (Cardiac disorders) | 1 (1) | 0 (0)
increased libido (Nervous system disorders) | 0 (0) | 1 (1)
coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
breast discharge (Endocrine disorders) | 0 (0) | 1 (1)
swollen lymph nodes (Immune system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small number of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No